CLINICAL TRIAL: NCT04612231
Title: Examining the Efficacy of the TEACCH School Transition to Employment and Post-Secondary Education Program
Brief Title: Examining the Efficacy of the T-STEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-0627; CDMRP-R180178-A (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2020-10-22; First posted 2020-11-02 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Autism Spectrum Disorder
Keywords: Transition; High-Functioning; Social Skills; Executive Functioning; Self-Advocacy; Higher Education; Career Exploration
MeSH Terms: conditions — Autism Spectrum Disorder; Social Skills | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: The statistician will use a random number generator to assign participants to the T-STEP Intervention condition or the Counseling Only Intervention condition. Assignment will be made separately at each site and with equal numbers assigned to each condition. This will ensure that equal numbers of participants are assigned to each condition across sites per year.
Masking Description: Research assistants will be masked to control for biases while administering the objective measure at baseline and post- assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T-STEP Intervention (Active Comparator): The T-STEP is a comprehensive 12-week transition program that will be delivered in a community college setting. The curriculum includes 36 hours of group-based instruction delivered within a traditional school academic semester (i.e., 24 ninety-minute classes across 12 weeks). Students also participate in a weekly community-based internship to practice the skills learned in the intervention group (2 hours per week for 12 weeks). In addition, students participate in 12 hours of manualized individual counseling services that are traditionally available on a college campus (e.g., job exploration/career counseling, academic counseling, and self-advocacy counseling).
  Interventions: Behavioral: TEACCH School Transition to Employment and Postsecondary Education (T-STEP)
- Counseling Only Intervention (Active Comparator): Participants in the Counseling Only condition will receive the same manualized counseling sessions that are included in the T-STEP program. Specifically, 12 hours of individual counseling focused on job exploration/career counseling, academic counseling, and self-advocacy counseling.
  Interventions: Behavioral: Counseling Services Alone

INTERVENTIONS:
Behavioral: TEACCH School Transition to Employment and Postsecondary Education (T-STEP) — The T-STEP Program is a 12-week transition intervention targeting specific challenges that young adults with ASD experience in executive function, social communication, and emotion regulation including group intervention, internship, and counseling services
  Arms: T-STEP Intervention
Behavioral: Counseling Services Alone — The Counseling Services Alone Intervention will receive 12 hours of individual counseling focused on job exploration/career counseling, academic counseling, and self-advocacy counseling.
  Arms: Counseling Only Intervention

SUMMARY:
The objective of this study is to evaluate the TEACCH School Transition to Employment and Post-Secondary Education (T-STEP) Program. Through randomized assignment young adults (18-21 year-old) with ASD will participate in the full T-STEP Program or a counseling only condition. Effectiveness will be assessed by caregiver report (social communication, executive function, employment readiness), self-report (self-determination, coping, depression), and behavioral observation (i.e., a mock employment experience). The long-term impact of this intervention is to promote a more positive quality of life for young adults with high functioning ASD including increased postsecondary education completion, employment, self-determination, and decreased difficulties with coping and depression.

DETAILED DESCRIPTION:
The purpose of the proposed study is to conduct an alternative treatment randomized clinical trial (RCT) to examine the efficacy of the TEACCH School Transition to Employment and Postsecondary Education (T-STEP) Program, a 12-week transition intervention targeting specific challenges that young adults with ASD experience in executive function, social communication, and emotion regulation including group intervention, internship, and counseling services, compared to counseling services only. The investigator predicts that the full T-STEP program (community college course, internship, counseling) will lead to improved short-term and long-term outcomes compared to counseling services only.

One cohort will be conducted per semester at two different community colleges with the specific semester counterbalanced across years. Each site will run one to two cohorts per year. The study will be conducted for three years. Students will be enrolled in the study after screening inclusion criteria have been met.

1. Screening. After contact, initial eligibility criteria will be confirmed during a phone screening documenting age, previous diagnosis of ASD, and completion, or in the final year of completing, a high school diploma.
2. Pre-Assessment. Young adults and caregivers will complete an assessment at their regional community college or via video visit (depending on COVID-19 restrictions) to verify eligibility. Following verification students will be randomized to the T-STEP Comprehensive intervention or the Counseling Only intervention.

   The statistician will use a random number generator to assign participants to the T-STEP Comprehensive intervention condition or the Counseling Only condition. The statistical consultant will use a random number generator to assign participants to the T-STEP Comprehensive intervention condition or the Counseling Only condition. Assignment will be made separately at each site and with equal numbers assigned to each condition. This will ensure that equal numbers of participants are assigned to each condition across sites per year.
3. Baseline. Baseline assessments are estimated to take 2 hours (1 hour for behavioral measures; 1 hour for self-report paper and pencil measures). Caregiver measures are estimated to take 1 to 1.5 hours. Assessments will take place on the community college campus or via video visit (depending on COVID-19 restrictions).
4. Intervention. Both treatment conditions will be offered free of charge through our partnership with participating community colleges. Participants in both groups will complete 12-weeks of treatment as described below. All sessions will occur at regional community college campuses via video sessions, or via a hybrid approach with some sessions virtually and some sessions on campus (depending on COVID-19 restrictions).

   T-STEP Intervention Condition. The T-STEP is a comprehensive 12-week transition program that will be delivered in a community college setting. The curriculum includes 36 hours of group-based instruction delivered within a traditional school academic semester (i.e., 24 ninety-minute classes across 12 weeks). Students also participate in a weekly community-based internship to practice the skills learned in the intervention group (2 hours per week for 12 weeks). In addition, students participate in 12 hours of manualized individual counseling services that are traditionally available on a college campus (e.g., job exploration/career counseling, academic counseling, and self-advocacy counseling).

   Counseling Only Intervention Condition. Participants in the Counseling Only condition will receive the same manualized counseling sessions that are included in the T-STEP program described above. Specifically, 12 hours of individual counseling focused on job exploration/career counseling, academic counseling, and self-advocacy counseling.
5. Post-Intervention (Post-Test) & Follow-Up. Participants in both conditions will complete post-assessments immediately following treatment and a follow-up assessment 4 months (week 28) after finishing the treatment. All assessments will take place on the community college campus or via video visit (depending on COVID-19 restrictions). Both assessments will take approximately 2 hours to complete by students with ASD and 35 minutes to complete by caregivers. Assessments will be completed by research assistants who are unfamiliar to participants.

ELIGIBILITY:
Inclusion Criteria:

* 16-21 years old
* Has completed (or in the final year of completing) a high school diploma
* Has a previous diagnosis of ASD to be confirmed by 1) an educational diagnosis of ASD as determined by a high school IEP for autism services; and/or (2) a psychological evaluation report
* Report documenting the diagnosis of ASD within the past 5 years
* Has a minimum Full-Scale IQ score of 80 as assessed by the Wechsler Abbreviated Scale of Intelligence-II
* Has a parent or other family member/surrogate who has regular contact with the young adult who will attend the assessment visit and report on the young adult's behaviors.
* English speaking.

Exclusion Criteria:

* Individuals younger than 16 or older than 21 years old
* No documentation of a previous Autism diagnosis
* Has a minimum Full-Scale IQ score less than 80 as assessed by the Wechsler Abbreviated
* The young adult does not have a family member/surrogate who can report on their behaviors.
* Non-English speaking

Ages: 16 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Change in Becker Work Adjustment Profile-2 (BWAP) Scores from Baseline to Post-Intervention | Baseline, post-intervention (within 4 weeks of completing the 12-week intervention)
  The BWAP is a 63-item informant report measure completed by the caregiver that evaluates skills important for job readiness and work performance across four domains: Work Habits/Attitudes, Interpersonal Relations, Cognitive Skills, and Work Performance Skills. T-Scores (27-73) for each domain will be calculated. A lower T-Score indicates more impairment on the given domain.
Change in Behavioral Rating Inventory of Executive Function, Adult Version (BRIEF-A) Scores from Baseline to Post-Intervention | Baseline, post-intervention (within 4 weeks of completing the 12-week intervention)
  The BRIEF-A is a 75-item informant report questionnaire that assesses a variety of behavioral manifestations of executive function (e.g., Inhibit, Self-Monitor, Plan/Organize, Shift, Initiate, Task Monitor, Emotional Control, Working Memory, and Organization of Materials) as well as a composite score of executive function. The informant report will be completed by the caregiver. T-Scores of subscales (Inhibit 39-88; Shift 38-84; Emotional Control 39-77; Self-Monitor 37-79; Initiate 36-83; Working Memory 39-90; Plan/Organize 38-83; Task Monitor 38-84; Organization of materials 37-75), Index scores (e.g., Behavioral Regulation 36-85; Metacognition 36-86) and the total score (e.g., Global Executive Composite 35-88) will be calculated. Lower T-Scores indicate higher levels of executive function and a better outcome.
Change in Transition Readiness and Employability Evaluation (TREE) Scores from Baseline to Post-Intervention | Baseline, post-intervention (within 4 weeks of completing the 12-week intervention)
  An objective behavioral observation measure developed that provides a series of organization, social communication, and emotion regulation presses during a simulated work environment appropriate for students with ASD and average or higher IQ. Two 15-minute employment tasks appropriate to office (e.g., filing, assembly of information folders) and computer data entry (e.g., accounting receipts, entry of evaluations forms) settings are presented. Participants have opportunities for social interaction with co-workers and supervisors, to respond to corrective feedback, and to request assistance. Assessments will be videotaped and coded by a trained research assistant who will be blind to treatment condition. Domain raw scores will be calculated (Emotion Regulation 0-16; Executive Function 0-16; Social Communication 0-22). Lower scores in each domain indicate less impairment and a better outcome.
Change in The American Institutes for Research Self-Determination Scale (AIR) Scores from Baseline to Post-Intervention | Baseline, post-intervention (within 4 weeks of completing the 12-week intervention)
  The AIR is a 24 item self-report measure, and an 18 item parent report of self-determination including a measure of knowledge and opportunity to modify and engage in events that affect the participant's wants and needs. The AIR's items are rated on a 5-point Likert scale. The Level of Self-Determination total raw score will be calculated for the self-report (0-120) and the parent report (0-90). A higher score indicates higher levels of self-determining behaviors and a better outcome.
Change in Coping Self-Efficacy Scale (CES) Scores from Baseline to Post-Intervention | Baseline, post-intervention (within 4 weeks of completing the 12-week intervention)
  The CSE is a 26-item self-report questionnaire completed by the student with ASD that measures an individual's confidence in using coping behaviors when faced with problems or life challenges. The CSE will be used to measure emotion regulation across three raw scored subscales (e.g., problem-focused coping, 0-48; stopping unpleasant emotions and thoughts, 0-36; and getting support from friends and family, 0-20) and the total raw score (0-104). A higher raw score indicates more self-confidence in an individual's ability to use coping behaviors and a better outcome.

SECONDARY OUTCOMES:
Change in Center for Epidemiological Studies - Depression, Revised (CESD-R) Scores | Up to 28 weeks
  The 20-item self-report version of the CESD-R, completed by the student with ASD, will be used to assess symptoms of depression. Respondents are asked to answer each question using a 4-point Likert scale from "less than one day" to "5-7 days" to describe their feelings (e.g., "I felt sad.") during the past week. The Total CESD-R Score will be calculated as a sum of responses to all 20 questions (0-60). A lower score indicates less depressive symptoms and a better outcome. Assessed at Baseline, post-intervention, and 4 month follow up.
Change in State Trait Anxiety Inventory (STAI) Trait Scale Scores | Up to 28 weeks
  A 20-item self-report completed by the student with ASD used to assess symptoms of anxiety. Respondents are asked to answer each question using a 4-point Likert scale from "almost never" to "almost always." The total score (20-80) will be used as a moderator of intervention efficacy and as an immediate outcome. A low score indicates less impairment of general anxiety and a better outcome. Assessed at Baseline, post-intervention, and 4 month follow up.
Student Adaptation to College Questionnaire (SACQ) | 4 month post-intervention completion follow up
  The SACQ is a self-report measure completed by the student with ASD of adjustment to college in four areas: Academic Adjustment, Social Adjustment, Personal-Emotional Adjustment, and Institutional Attachment. T-Scores will be calculated for the four domains and the total score (25-75). Conversion tables are categorized by gender and year in college. Higher scores indicates better adjustment to college and a better outcome.
Change in Grade Point Average (GPA) | Baseline, 4 month post-intervention completion follow up, a total of up to 28 weeks
  GPA will be collected to measure change in success following completion of the intervention. Better outcomes are indicated by increased GPA.
Change in Employment Status Categorizations | Baseline, 4 month post-intervention completion follow up, a total of up to 28 weeks
  Employment status will be measured through quantitative categorizations of employment wages (e.g., under minimum wage, minimum wage, above minimum wage, unpaid volunteer; 1-4) and number of hours worked per week (e.g., less than 5 hours, 5-9 hours, 10-19 hours, 20-29 hours, 30-29 hours, 40 hours; 1-6). Maintenance or increase of employment wages and number of hours worked per week is a better outcome.
Change in Becker Work Adjustment Profile-2 (BWAP) Scores from Post-Intervention to 4 Month Follow Up | Post-Intervention (within 4 weeks of completing the 12-week intervention), 4 month post-intervention completion follow up, a total of up to 16 weeks
  The BWAP is a 63-item informant report measure completed by the caregiver that evaluates skills important for job readiness and work performance across four domains: Work Habits/Attitudes, Interpersonal Relations, Cognitive Skills, and Work Performance Skills. T-Scores (27-73) for each domain will be calculated. A lower T-Score indicates more impairment on the given domain.
Change in Behavioral Rating Inventory of Executive Function, Adult Version (BRIEF-A) Scores from Post-Intervention to 4 Month Follow Up | Post-Intervention (within 4 weeks of completing the 12-week intervention), 4 month post-intervention completion follow up, a total of up to 16 weeks
  The BRIEF-A is a 75-item informant report questionnaire that assesses a variety of behavioral manifestations of executive function (e.g., Inhibit, Self-Monitor, Plan/Organize, Shift, Initiate, Task Monitor, Emotional Control, Working Memory, and Organization of Materials) as well as a composite score of executive function. The informant report will be completed by the caregiver. T-Scores of subscales (Inhibit 39-88; Shift 38-84; Emotional Control 39-77; Self-Monitor 37-79; Initiate 36-83; Working Memory 39-90; Plan/Organize 38-83; Task Monitor 38-84; Organization of materials 37-75), Index scores (e.g., Behavioral Regulation 36-85; Metacognition 36-86) and the total score (e.g., Global Executive Composite 35-88) will be calculated. Lower T-Scores indicate higher levels of executive function and a better outcome.
Change in The American Institutes for Research Self-Determination Scale (AIR) Scores from Post-Intervention to 4 Month Follow Up | Post-Intervention (within 4 weeks of completing the 12-week intervention), 4 month post-intervention completion follow up, a total of up to 16 weeks
  The AIR is a 24 item self-report measure, and an 18 item parent report of self-determination including a measure of knowledge and opportunity to modify and engage in events that affect the participant's wants and needs. The AIR's items are rated on a 5-point Likert scale. The Level of Self-Determination total raw score will be calculated for the self-report (0-120) and the parent report (0-90). A higher score indicates higher levels of self-determining behaviors and a better outcome.
Change in Coping Self-Efficacy Scale (CES) Scores from Post-Intervention to 4 Month Follow Up | Post-Intervention (within 4 weeks of completing the 12-week intervention), 4 month post-intervention completion follow up, a total of up to 16 weeks
  The CSE is a 26-item self-report questionnaire completed by the student with ASD that measures an individual's confidence in using coping behaviors when faced with problems or life challenges. The CSE will be used to measure emotion regulation across three raw scored subscales (e.g., problem-focused coping, 0-48; stopping unpleasant emotions and thoughts, 0-36; and getting support from friends and family, 0-20) and the total raw score (0-104). A higher raw score indicates more self-confidence in an individual's ability to use coping behaviors and a better outcome.
Change in Activities of Daily Living (WADL) Scores | Up to 28 weeks
  The WADL is a 17-item informant report questionnaire that assesses current levels of independence in performing activities of daily living. Respondents are asked to answer each question using a 3-point Likert scale from "does not do at all" to "independent/does on own" to describe the person's level of independence. The Total WADL Score will be calculated as a sum of responses to all 17 questions (0-34). A higher score indicates more independence and a better outcome. Assessed at Baseline, post-intervention, and 4-month follow-up.
Change in Clinical Global Impression Scale (CGI) Scores from Baseline to Post-Intervention | Baseline, post-intervention (within 4 weeks of completing the 12-week intervention)
  The CGI is completed by the interventionist and assesses transition readiness on a 7-point scale. Higher scores correspond to better transition readiness.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Klinger, Ph.D., Principal Investigator — University of North Carolina, Chapel Hill; Brianne Tomaszewski, Ph.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (5):
- United States (5):
  - University of North Carolina, Chapel Hill, North Carolina
  - Johnston Community College, Clayton, North Carolina
  - Alamance Community College, Graham, North Carolina
  - Guilford Technical Community College, Greensboro, North Carolina
  - Wake Tech Community College, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared via the National Database for Autism Research (NDAR). In addition, an NDAR study for each publication that underlies results of the study will be created so that readers of the article can link back to the data used in NDAR.
Supporting Information: Study Protocol
Time Frame: Descriptive/raw deidentified data will be reported semi-annually through NDAR. Other experimental data will be shared after the primary objectives of the study have been met.
Access Criteria: Request login access to NDAR data
URL: http://ndar.nih.gov

DOCUMENTS (1):
  • Informed Consent Form (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/31/NCT04612231/ICF_000.pdf